CLINICAL TRIAL: NCT01086553
Title: Double-blind, Double-dummy, Randomised, Comparative, Multi-centre Phase III Study on the Efficacy and Tolerability of an 8-week Oral Treatment With 9 mg Budesonide Once Daily vs. 3 mg Budesonide Three-times Daily in Patients With Active Crohn's Disease
Brief Title: 9 mg Budesonide Once Daily (OD) Versus 3 mg Budesonide Three Times Daily (TID) in Active Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUG-2/CDA; 2008-006957-42 (EudraCT Number)
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Crohn´s Disease
Keywords: Crohn´s disease; budesonide; induction of remission
MeSH Terms: conditions — Crohn Disease | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): 9mg budesonide OD
  Interventions: Drug: budesonide
- B (Active Comparator): 3mg budesonide TID
  Interventions: Drug: budesonide

INTERVENTIONS:
Drug: budesonide — 9mg budesonide OD
  Arms: A
Drug: budesonide — 3mg budesonide TID
  Arms: B

SUMMARY:
This study aims to evaluate the efficacy of 9 mg budesonide once daily (OD) versus 3 mg budesonide three-times daily (TID) for the induction of remission in Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* Age 18 to 75 years,
* Symptoms of Crohn's disease since at least 3 months; diagnosis confirmed by endoscopic and histological, or endoscopic and radiological criteria [endoscopy not older than 12 months or if older, then clinical signs (e.g., pain localisation, pain intensity, blood in stool) and behaviour (according to Montreal classification) should be unchanged compared to former episodes],
* Localisation of CD either in terminal ileum, coecum, ascending colon, or ileocolitis,
* Active phase of disease (200 < CDAI < 400),
* Negative pregnancy test in females of childbearing potential,
* Women of child-bearing potential have to apply appropriate contraceptive methods, e.g., hormonal contraception, intrauterine device (IUD), double-barrier method of contraception (e.g., use of a condom and spermicide), or partner has undergone vasectomy. The investigator is responsible for determining whether the subject has adequate birth control for study participation.

Exclusion Criteria:

* Known Crohn's lesions in the upper GI-tract (up to and including the jejunum) or rectum with present symptoms,
* Septic complications,
* Evidence of infectious diarrhoea (i.e., pathogenic bacteria in stool culture),
* Abscess, perforation, or active fistulas,
* Ileostomy or colostomy,
* Resection of more than 50 cm of the ileum,
* Bowel surgery within the last 3 months,
* Immediate surgery required (e.g., major stenosis, serious bleeding, peritonitis, ileus),
* Clinical signs of stricturing disease,
* Subileus within the last 6 months (subileus with inflammatory hint allowed),
* Suspicion of ileus, subileus or corresponding symptoms,
* Parenteral or tube feeding,
* Active peptic ulcer disease, local intestinal infection, or known established cataract,
* Diabetes mellitus, infection, osteoporosis, glaucoma, tuberculosis, or hypertension if careful medical monitoring is not ensured,
* Abnormal hepatic function (ALT or ALP > 2.5 x upper limit of normal [ULN]), liver cirrhosis, or portal hypertension,
* Abnormal renal function (Cystatin C > ULN),
* Any severe concomitant cardiovascular, renal, endocrine, or psychiatric disorder,
* History of cancer in the last five years (except for non-metastatic cancers, e.g., basalioma),
* Treatment with immunosuppressants or anti-cancer drugs, e.g., 6 TG, methotrexate, tacrolimus, cyclophosphamide, or cyclosporine within the last 3 months; in case of treatment with azathioprine or 6 MP the drugs have to be used for maintenance of remission only and dosage has to be unchanged within the last 3 months before baseline visit and during the study,
* Treatment with ketoconazole or other CYP3A inhibitors within the last month before baseline visit,
* Treatment with anti-TNF-alpha therapy within 3 months before baseline visit,
* Conventional steroids (iv, po, rectal) within 2 weeks before baseline visit,
* > 6 mg/d budesonide po within 2 weeks before baseline visit,
* Steroids for inhalation within 2 weeks before baseline visit,
* Patients known to be steroid-refractory,
* Treatment of study disease with oral antibiotics (e.g., metronidazole or ciprofloxacin) within the last 2 weeks,
* Application of non-steroidal anti-inflammatory drugs (NSAIDs) within 2 weeks before baseline visit except ≤ 350 mg/d or short-term acetylsalicylic acid (paracetamol is allowed),
* Known intolerance/hypersensitivity to study drug,
* Well-founded doubt about the patient's cooperation, e.g., because of addiction to alcohol or drugs,
* Existing or intended pregnancy or breast-feeding,
* Participation in another clinical trial within the last 30 days, simultaneous participation in another clinical trial, or previous participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Rate of clinical remission, defined as a CDAI < 150, at week 8 (LOCF) | 8 weeks

SECONDARY OUTCOMES:
Response to treatment defined as CDAI < 150 or CDAI reduction of > 100 points | 8 weeks
Adverse events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Axel Dignass, Prof., Principal Investigator — Med. Klinik I - Markus-Krankenhaus - Frankfurter Diakonie-Kliniken
Locations (1):
- Med. Klinik I - Markus-Krankenhaus - Frankfurter Diakonie-Kliniken, Frankfurt, Germany

REFERENCES:
- [Result] Dignass A, Stoynov S, Dorofeyev AE, Grigorieva GA, Tomsova E, Altorjay I, Tuculanu D, Bunganic I, Pokrotnieks J, Kupcinskas L, Dilger K, Greinwald R, Mueller R; International Budenofalk Study Group. Once versus three times daily dosing of oral budesonide for active Crohn's disease: a double-blind, double-dummy, randomised trial. J Crohns Colitis. 2014 Sep;8(9):970-80. doi: 10.1016/j.crohns.2014.01.021. Epub 2014 Feb 15. PMID 24534142